CLINICAL TRIAL: NCT02875067
Title: A Phase I/II Study of the Combination of Pembrolizumab and Lenalidomide, in Patients With Relapsed Non-Hodgkin and Hodgkin Lymphoma
Brief Title: Safety & Efficacy Study of Combination of Pembrolizumab and Lenalidomide, in Patients With Relapsed Non-Hodgkin and Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Merck's decision for early termination of the data
Sponsor: NYU Langone Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-00285
Record Dates: First submitted 2016-08-08; First posted 2016-08-23 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Relapsed Hodgkin Lymphoma; Relapsed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — pembrolizumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and Lenalidomide (Experimental): An intravenous infusion of 200 mg of pembrolizumab (MK3475) once every 3 weeks for a total of 4 infusions
  Lenalidomide at either 15 mg, 10 mg or 20 mg (depending on which cohort patients are enrolled in) days 1-14 every 21 days
  Interventions: Biological: Pembrolizumab; Drug: Lenalidomide

INTERVENTIONS:
Biological: Pembrolizumab
  Other Names: MK3475; Keytruda
Drug: Lenalidomide
  Other Names: Revlimid

SUMMARY:
This trial is to assess the safety & efficacy of the Combination of Pembrolizumab and Lenalidomide in the management of patients with Relapsed Hodgkin Lymphoma.

DETAILED DESCRIPTION:
There is an emerging clinical data to confirm that Programmed death-1 (PD-1)blockade is safe and viable in lymphoma.

The investigators hypothesize that the novel immune platform of pembrolizumab and lenalidomide, will be safe and well tolerated in patients with Relapsed Refractory (RR) Hodgkin Lymphoma (HL) and non-Hodgkin lymphoma (NHL) and that this combination will result in a complete response (CR) rate of 50% in patients with RR HL.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Have measurable or evaluable disease, as defined in 2007 Revised Response Criteria for Malignant Lymphoma24 and have received at least two prior therapies. HL patients must not be currently eligible for autologous stem cell transplant.
4. Be willing to provide either archived tumor tissue or tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1.
5. Have a performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
6. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 14 days of treatment initiation.

   Adequate Organ Function Laboratory Values:
   * Absolute neutrophil count (ANC): ≥1,000 /microliter (mcL)
   * Platelets: ≥75,000 / mcL
   * Hemoglobin: ≥9 g/dL or ≥5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
   * Serum creatinine OR: ≤1.5 X upper limit of normal (ULN) OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl): ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
   * Serum total bilirubin: ≤ 1.5 X ULN OR
   * Direct bilirubin ≤ ULN for subjects with total bilirubin levels: >1.5 ULN
   * Aspartate aminotransferase (AST) / serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/ serum glutamic pyruvic transaminase (SGPT): ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
   * Albumin: >2.5 mg/dL
   * International Normalized Ratio (INR) or Prothrombin Time (PT): ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
   * Activated Partial Thromboplastin Time (aPTT): ≤1.5 X ULN unless subject is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants

   aCreatinine clearance should be calculated per institutional standard.
7. Female subject of childbearing potential should have two negative urine or serum pregnancy test, one at 10-14 days before first dose of study drug and another within 24 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
9. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active Bacillus Tuberculosis (TB)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C virus (HCV) (e.g., HCV Ribonucleic acid (RNA) [qualitative] is detected), or other active viral hepatitis. Patients with treated and resolved hepatitis B or C are eligible. Patients with active liver disease, except liver abnormalities directly attributable to lymphoma are ineligible,
18. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Diefenbach, MD, Principal Investigator — NYU Perlmutter Cancer Center
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - NYU Perlmutter Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab and Lenalidomide: An intravenous infusion of 200 mg of pembrolizumab (MK3475) once every 3 weeks for a total of 4 infusions
  Lenalidomide at either 15 mg, 10 mg or 20 mg (depending on which cohort patients are enrolled in) days 1-14 every 21 days
  Pembrolizumab
  Lenalidomide
Period: Overall Study
Arm/Group | Pembrolizumab and Lenalidomide
Started | 6
Completed | 0
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Withdrawal by Termination of Study | 5

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab and Lenalidomide
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Assess Safety and Tolerability of the Combination of Pembrolizumab and Lenalidomide (Number of Drug Related Adverse Events)
Description: Assessing the number of drug related adverse events at each dose level of lenalidomide
Time Frame: up to 2 years
Population: The study was terminated before formal data collection could occur.
Arm/Group | Pembrolizumab and Lenalidomide
Number analyzed (Participants) | 0

2. Primary Outcome: Estimate Overall Response Rate (ORR)
Description: Assessment of lymphoma response (CR, PR or SD) and disease progression will be evaluated according to the Revised Response Criteria for Malignant Lymphoma. Overall response will be measured for all patients who complete one cycle of treatment
Time Frame: up to 2 years
Population: The study was terminated before formal data collection could occur.
Arm/Group | Pembrolizumab and Lenalidomide
Number analyzed (Participants) | 0

3. Primary Outcome: Estimate Complete Response Rate (CR)
Description: as for outcome 2
Time Frame: up to 2 years
Population: The study was terminated before formal data collection could occur.
Arm/Group | Pembrolizumab and Lenalidomide
Number analyzed (Participants) | 0

4. Primary Outcome: Estimate Partial Response Rate (PR)
Description: as for outcome 2
Time Frame: up to 2 years
Population: The study was terminated before formal data collection could occur.
Arm/Group | Pembrolizumab and Lenalidomide
Number analyzed (Participants) | 0

5. Secondary Outcome: Estimate the ORR (CR, PR) for Combination Within & Across Dose Levels of Lenalidomide
Description: as for outcome 2
Time Frame: up to 2 years
Population: The study was terminated before formal data collection could occur.
Arm/Group | Pembrolizumab and Lenalidomide
Number analyzed (Participants) | 0

6. Secondary Outcome: Estimate Stable Disease (SD) for Combination Within & Across Dose Levels of Lenalidomide
Description: Assessment of lymphoma response (CR, PR or SD) and disease progression will be evaluated according to the Revised Response Criteria for Malignant Lymphoma. Overall response will be measured for all patients who complete one cycle of treatment. Kaplan-Meir methodology will be used to estimate median PFS and Overall Survival (OS).
Time Frame: up to 2 years
Population: The study was terminated before formal data collection could occur.
Arm/Group | Pembrolizumab and Lenalidomide
Number analyzed (Participants) | 0

7. Secondary Outcome: Estimate Progression Free Survival (PFS) for Combination Within & Across Dose Levels of Lenalidomide
Description: Assessment of lymphoma response (CR, PR or SD) and disease progression will be evaluated according to the Revised Response Criteria for Malignant Lymphoma. Overall response will be measured for all patients who complete one cycle of treatment. Kaplan-Meir methodology will be used to estimate median PFS and OS.
Time Frame: up to 2 years
Population: The study was terminated before formal data collection could occur.
Arm/Group | Pembrolizumab and Lenalidomide
Number analyzed (Participants) | 0

8. Secondary Outcome: Estimate Clinical Benefit (Including SD) for the Combination
Description: as for outcome 7
Time Frame: up to 2 years
Population: The study was terminated before formal data collection could occur.
Arm/Group | Pembrolizumab and Lenalidomide
Number analyzed (Participants) | 0

9. Secondary Outcome: Estimate Progression Free Survival (PFS) for the Combination
Description: as for outcome 7
Time Frame: up to 2 years
Population: The study was terminated before formal data collection could occur.
Arm/Group | Pembrolizumab and Lenalidomide
Number analyzed (Participants) | 0

10. Secondary Outcome: Estimate Duration of Response (DOR) for the Combination
Description: as for outcome 7
Time Frame: up to 2 years
Population: The study was terminated before formal data collection could occur.
Arm/Group | Pembrolizumab and Lenalidomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The study was terminated before formal data collection could occur.
Arm/Group | Pembrolizumab and Lenalidomide
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT02875067/Prot_SAP_000.pdf